CLINICAL TRIAL: NCT02251769
Title: A Single-centre Open-label Study in Healthy Adult Volunteers to Determine the Effects of Single-dose and Steady-state TPV/r (500 mg/200 mg) on the Steady-state Pharmacokinetics of Clarithromycin (BIAXIN®) 500 mg Bid and a Preliminary Assessment of the Effects of a Standard High-fat Test Meal on the Steady-state Pharmacokinetics of Tipranavir
Brief Title: Effects of Single-dose and Steady-state TPV/r on the Steady-state Pharmacokinetics of Clarithromycin and a Preliminary Assessment of the Effects of a Standard High-fat Test Meal on the Steady-state Pharmacokinetics of Tipranavir
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1182.11
Record Dates: First submitted 2014-09-25; First posted 2014-09-29 (Estimated); Last update posted 2014-09-29 (Estimated); Status verified 2014-09

CONDITIONS: Healthy
MeSH Terms: interventions — tipranavir; Ritonavir; Clarithromycin

ARMS (1):
- Sequential administration (Experimental)
  Interventions: Drug: Tipranavir; Drug: Ritonavir; Drug: Clarithromycin; Other: High-Fat Test Meal

INTERVENTIONS:
Drug: Tipranavir
Drug: Ritonavir
Drug: Clarithromycin
Other: High-Fat Test Meal

SUMMARY:
To determine the effects of single-dose and steady-state Tipranavir/Ritonavir (TPV/r) at 500 mg/200 mg bid on the steady-state pharmacokinetics of clarithromycin and to determine the effects of a standard high-fat test meal on the steady-state pharmacokinetics of tipranavir.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects between 18 and 60 years of age inclusive
* A Body Mass Index (BMI) between 18 and 29 kg/m2
* Signed informed consent prior to trial participation
* Ability to swallow multiple capsules without difficulty
* Ability to ingest a standard high-fat test meal
* Acceptable laboratory values that indicated adequate baseline organ function were required at the time of screening. Laboratory values were considered to be acceptable if severity was less than or equal to Grade 1, based on the AIDS Clinical Trials Group (ACTG) Grading Scale
* Acceptable medical history, physical examination and 12-lead ECG were required prior to entering the treatment phase of the study
* Willingness to abstain from alcohol for 48 hours prior to study Day 0 and abstain from alcohol for the duration of the study. In addition, ingestion of red wine is not allowed within 5 days prior to Day 0 (Visit 2)
* Willingness to abstain from grapefruit or grapefruit juice or products containing grapefruit juice starting 10 days prior to any administration of study drug up until the end of the study
* Willingness to abstain from ingestion of Seville oranges, garlic supplements, St. John's Wort, or Milk Thistle, within 5 days of treatment and for the duration of the study
* Willingness to abstain from methylxanthine-containing drinks or foods (coffee, tea, cola, energy drinks, chocolate, etc.) within 48 hours of each pharmacokinetic sampling day and until after the last sample from each of the intensive sampling days was collected
* Willingness to abstain from over the counter herbal medications for the duration of the study
* Willingness to abstain from vigorous physical exercise during intensive pharmacokinetic days
* Reasonable probability for completion of the study
* Non-smokers for at least 3 months prior to Day 0

Exclusion Criteria:

* Female subjects who are of reproductive potential and who:

  1. Have positive serum β-hCG at Visit 1, or on Day 0
  2. Are not using a barrier contraceptive method for at least 3 months prior to Visit 2 (Day 0)
  3. Are not willing to use a reliable method of barrier contraception (such as diaphragm or condoms), during the trial and for 30 days after trial completion/termination
  4. Are breast-feeding
* Use of any pharmacological contraceptive (including oral, patch or injectable contraceptives) within 1 month prior to study initiation and for the duration of the study
* Use of hormone replacement therapy within 1 month prior to study initiation and for the duration of the study
* Participation in another trial with an investigational medicine within 60 days prior to Day 0 (Visit 2)
* Use of any prohibited medication listed in the protocol within 30 days prior to Day 0 (Visit 2)
* Administration of antibiotics within 10 days prior to Day 0 (Visit 2) or during the trial
* History of acute illness within 60 days of trial initiation. Subjects are excluded for these disorders greater than 60 days if, in the opinion of the investigator, the subject does not qualify as a healthy volunteer
* Serological evidence of hepatitis B (HBV) or hepatitis C (HCV)
* Serological evidence of exposure to HIV
* Recent history of alcohol or substance abuse (within 6 months of study period)
* Blood or plasma donations within 30 days prior to Day 0 (Visit 2) or during the trial
* Subjects with a seated systolic blood pressure either <100 mm Hg or >150 mm Hg
* Subjects with a history of any illness or allergy that, in the opinion of the investigator, might confound the results of the study or pose additional risk in administering tipranavir (TPV), ritonavir (RTV) or clarithromycin (CLR) to the subject
* Subjects who have taken, within 7 days prior to Day 0 (Visit 2), any over-the-counter or prescription drugs that, in the opinion of the investigator in consultation with the BI clinical monitor, might interfere with either the absorption, distribution or metabolism of the test substances
* Known hypersensitivity to TPV, RTV, sulfonamides, or CLR
* Lactose intolerance or intolerance to high-fat foods
* Allergies or intolerance to foods such as soybean, wheat, milk, eggs or gluten
* Inability to adhere to requirements of the protocol

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2003-08; Primary Completion 2003-09 (Actual)

PRIMARY OUTCOMES:
Area under plasma concentration time curve from 0-12 hours (AUC0-12h) | up to 12 hours
Maximum plasma concentration (Cmax) | up to 12 hours
Plasma trough concentration (Cp12h) | up to 12 hours

SECONDARY OUTCOMES:
Oral clearance (CL/F) | up to 12 hours
Volume of distribution (V) | up to 12 hours
Apparent terminal half life (t1/2) | up to 12 hours
Time of maximum concentration (Tmax) | up to 12 hours
Mean Residency Time (MRT) | up to 12 hours
Number of patients with adverse events | up to day 13
Number of patients with clinically significant laboratory findings | up to day 13